CLINICAL TRIAL: NCT00392171
Title: The Temozolomide RESCUE Study: A Phase II Trial of Continuous (28/28) Dose-intense Temozolomide (CDIT) Chemotherapy After Progression on Conventional 5/28 Day Temozolomide in Patients With Recurrent Malignant Glioma
Brief Title: The Effects of Continuous 28-day (28/28) Temozolomide Chemotherapy in Subjects With Recurrent Malignant Glioma Who Have Failed the Conventional 5-day (5/28) Treatment (P04601)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04601
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — Temozolomide

ARMS (1):
- Temozolomide (Experimental): Temozolomide will be administered at a dose of 50 mg/m^2 for cycles of 28 days for 12 months or until progression.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Subjects will receive temozolomide 50 mg/m^2 for cycles of 28 days for 12 months or until progression
  Other Names: SCH 52365

SUMMARY:
The purpose of this non-randomized, open-label, multicenter, Phase II, 2-stage design, RESCUE study is to test the hypothesis that continuous 28-day oral dosing (28/28) with dose-intense temozolomide (50 mg/m^2) for up to 12 months may overcome resistance and be effective in the management of adult patients with malignant glioma who have failed following at least 2 cycles (2 months) of conventional 5-day (5/28) cycles of high-dose temozolomide (150-200 mg/m^2).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, greater than 18 years old.
* Surgically confirmed diagnosis of malignant glioma, specifically anaplastic glioma (anaplastic astrocytoma [AA], anaplastic oligodendroglioma [AO], anaplastic oligoastrocytoma [AOA]) or glioblastoma multiforme (GBM).
* Must have completed at least 2 cycles (2 months) of conventional 5/28 temozolomide, with radiological evidence of progression.
* GBM treated with concurrent chemoradiation with temozolomide according to the EORTC/NCIC (European Organization for Research & Treatment of Cancer/National Cancer Institute of Canada) protocol.
* Evidence of progression confirmed radiologically (CT [computed tomography] or MRI [magnetic resonance imaging]).
* Patients must be enrolled within 2 weeks of last radiological confirmation of progression, except for patients undergoing surgical resection.
* Patients undergoing surgical resection for recurrent disease must be enrolled within 2 weeks of the post-surgical scan.
* Patients with no residual disease after surgery are allowed.
* Steroids dose should have been stabilized during the last 2 weeks prior to enrollment.
* Use of medically approved contraception in fertile males and females.
* Women of childbearing potential must have a negative urine or serum pregnancy test (urinary excretion or serum level of bHCG [beta human chorionic gonadotropin]) within 24 hours of inclusion in the study.
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
* Signed informed consent form.

Exclusion Criteria:

* GBM progression during the first 2 months of adjuvant temozolomide (5/28).
* AA progression during the first 2 months of standard temozolomide therapy (5/28).
* Chemotherapy for the malignant glioma other than temozolomide.
* More than one prior course of chemotherapy with temozolomide.
* Patient evolving from anaplastic glioma to GBM following primary therapy.
* Patient older than 70 years or who received no conventional chemoradiation regimen.
* Patient who received radiotherapy for recurrent disease.
* Patient with metastatic disease.
* Known human immunodeficiency virus (HIV) infection.
* History of non-compliance to other therapies.
* Inadequate hematological, renal and hepatic function according to all of the following laboratory values (to be performed within 14 days, inclusive, prior to study inclusion):
* Absolute neutrophil count <=1.5 ×10^9/L;
* Platelets <=100 ×10^9/L;
* Hemoglobin <90 g/L;
* Serum creatinine >=1.5 times upper limit of laboratory normal (ULN);
* Total serum bilirubin >=1.5 times ULN;
* ASAT (AST [aspartate aminotransferase]) or ALAT (ALT [alanine aminotransferase) >2.0 times ULN;
* Alkaline phosphatase of >2.5 times ULN.
* Known chronic hepatitis B or hepatitis C infection.
* Any other serious medical condition, according to the medical judgment of the physician prior to inclusion in the study.
* Any medical condition that could interfere with oral medication intake (e.g., frequent vomiting, partial bowel obstruction).
* Other malignancies during the previous 5 years with the exception of surgically cured carcinoma in-situ of the cervix and basal cell carcinoma or non-melanoma skin cancer.
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule as discussed with the patient before inclusion in the study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-06-09 (Actual); Primary Completion 2009-09-15 (Actual); Study Completion 2009-09-15 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Perry JR, Belanger K, Mason WP, Fulton D, Kavan P, Easaw J, Shields C, Kirby S, Macdonald DR, Eisenstat DD, Thiessen B, Forsyth P, Pouliot JF. Phase II trial of continuous dose-intense temozolomide in recurrent malignant glioma: RESCUE study. J Clin Oncol. 2010 Apr 20;28(12):2051-7. doi: 10.1200/JCO.2009.26.5520. Epub 2010 Mar 22. PMID 20308655

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide
Started | 120
Completed | 15
Not Completed | 105
Not completed — Did not meet inclusion criteria | 4
Not completed — Disease progression | 101

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 76
Region of Enrollment [Number; unit: participants]
  Canada | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Surviving at Six Months of Treatment Without Evidence of Disease Progression.
Description: Progression-free survival as determined by Kaplan-Meier method.
Time Frame: 6 months
Population: Participants who received allocated intervention.
  The percentage of participants reported is based on the number of participants within each category (not total number of all categories combined).
Measure: Number; unit: Percentage of Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 116
Percentage of Participants
  Anaplastic Glioma (n=28) | 35.7
  Early Glioblastoma Multiforme (GBM) (n=33) | 27.3
  Extended Glioblastoma Multiforme (GBM) (n=27) | 7.4
  Rechallenge Glioblastoma Multiforme (GBM) (n=28) | 35.7

ADVERSE EVENTS:
Arm/Group | Temozolomide
Serious Adverse Events (participants affected / at risk) | 27/120
Other Adverse Events (participants affected / at risk) | 111/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=120)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2)
IRRITABILITY (General disorders) | 1 (1)
PAIN (General disorders) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (2)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (2)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
APHASIA (Nervous system disorders) | 2 (2)
ATAXIA (Nervous system disorders) | 1 (1)
BALANCE DISORDER (Nervous system disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 4 (4)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1)
GRAND MAL CONVULSION (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2)
HEMIPARESIS (Nervous system disorders) | 1 (1)
HEMIPLEGIA (Nervous system disorders) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 1 (1)
MONOPARESIS (Nervous system disorders) | 1 (1)
POSTICTAL PARALYSIS (Nervous system disorders) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SPEECH DISORDER (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 3 (3)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=120)
NEUTROPENIA (Blood and lymphatic system disorders) | 7 (7)
VISION BLURRED (Eye disorders) | 7 (8)
CONSTIPATION (Gastrointestinal disorders) | 15 (16)
DIARRHOEA (Gastrointestinal disorders) | 8 (9)
DYSPEPSIA (Gastrointestinal disorders) | 7 (7)
NAUSEA (Gastrointestinal disorders) | 35 (40)
VOMITING (Gastrointestinal disorders) | 24 (29)
ASTHENIA (General disorders) | 8 (9)
FATIGUE (General disorders) | 48 (64)
GAIT DISTURBANCE (General disorders) | 13 (18)
OEDEMA (General disorders) | 7 (10)
OEDEMA PERIPHERAL (General disorders) | 9 (10)
ORAL CANDIDIASIS (Infections and infestations) | 10 (12)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (8)
BALANCE DISORDER (Nervous system disorders) | 9 (11)
CONVULSION (Nervous system disorders) | 16 (22)
DIZZINESS (Nervous system disorders) | 8 (11)
HEADACHE (Nervous system disorders) | 34 (51)
HEMIANOPIA (Nervous system disorders) | 8 (9)
HEMIPARESIS (Nervous system disorders) | 22 (31)
HYPOAESTHESIA (Nervous system disorders) | 7 (8)
MEMORY IMPAIRMENT (Nervous system disorders) | 17 (28)
MONOPARESIS (Nervous system disorders) | 11 (19)
SOMNOLENCE (Nervous system disorders) | 10 (12)
SPEECH DISORDER (Nervous system disorders) | 7 (9)
CONFUSIONAL STATE (Psychiatric disorders) | 13 (20)
INSOMNIA (Psychiatric disorders) | 13 (15)
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (16)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 (10)
RASH (Skin and subcutaneous tissue disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Chair agrees not to publish/present any interim results without prior Sponsor written consent. Investigators agree to provide 30 days to review prior to submission. Sponsor shall have proper representation/editorial rights/right to review/comment with regard to proprietary information. If the parties disagree concerning the appropriateness and/or confidentiality of information, Investigators agree to discuss and resolve any such issues prior to submission.